CLINICAL TRIAL: NCT05050864
Title: Randomized Controlled Trial Evaluating the Efficacy of Venous Sinus Stenting Versus Neurosurgical Internal Ventricular Shunt on Papillary Edema in the Management of Idiopathic Intracranial Hypertension
Brief Title: Stenting Versus Neurosurgical Treatment of Idiopathic Intracranial Hypertension.
Acronym: HYDROPTIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PBN_2021_4
Record Dates: First submitted 2021-09-10; First posted 2021-09-21 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Pseudotumor Cerebri; Cerebrospinal Fluid; Transverse Sinuses
Keywords: Endovacascular; ventricular shunt; papillary edema; visual field
MeSH Terms: conditions — Pseudotumor Cerebri

STUDY DESIGN:
Intervention Model Description: Name : internal ventricular shunt (neurosurgery)
  Description :
  The internal ventricular shunt consists of the introduction of a catheter from a lateral ventricle into the atrium or peritoneum. It is associated with a valve whose opening pressure is adjustable. The goal is that cerebrospinal fluid can be absorbed extra-cranial.
  Intervention 2 Name : endovacascular stenting (interventional neuroradiology)
  Description
  The placement of a vascular endoprosthesis (stent) is an interventional neuroradiology procedure aimed, by venous approach (percutaneous puncture), to restore the diameter of a venous sinus. It requires 6 months of antiplatelet aggregation. The aim is to allow better vscription : enous drainage from the brain to increase the absorption of cerebrospinal fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- internal ventricular shunt (neurosurgery) (Active Comparator): The internal ventricular shunt consists of the introduction of a catheter from a lateral ventricle into the atrium or peritoneum. It is associated with a valve whose opening pressure is adjustable. The goal is that cerebrospinal fluid can be absorbed extra-cranial
  Interventions: Procedure: Neurosurgical internal ventricular shunt
- endovacascular stenting (interventional neuroradiology) (Active Comparator): The placement of a vascular endoprosthesis (stent) is an interventional neuroradiology procedure aimed, by venous approach (percutaneous puncture), to restore the diameter of a venous sinus. It requires 6 months of antiplatelet aggregation. The aim is to allow better venous drainage from the brain to increase the absorption of cerebrospinal fluid.
  Interventions: Procedure: venous sinus stenting

INTERVENTIONS:
Procedure: venous sinus stenting — The placement of a vascular endoprosthesis (stent) is an interventional neuroradiology procedure aimed, by venous approach (percutaneous puncture), to restore the diameter of a venous sinus. It requires 6 months of antiplatelet aggregation. The aim is to allow better venous drainage from the brain to increase the absorption of cerebrospinal fluid
  Arms: endovacascular stenting (interventional neuroradiology)
Procedure: Neurosurgical internal ventricular shunt — The internal ventricular shunt consists of the introduction of a catheter from a lateral ventricle into the atrium or peritoneum. It is associated with a valve whose opening pressure is adjustable. The goal is that cerebrospinal fluid can be absorbed extra-cranial
  Arms: internal ventricular shunt (neurosurgery)

SUMMARY:
Idiopathic intracranial hypertension (HTICi) is a pathology, affecting young adults with a predominance of women, due to an increase in intracranial pressure, which may be associated with stenosis of the cerebral venous sinuses and whose origin remains unknown.

This hypertension can lead to papillary edema (OP) which can lead to a narrowing of the visual field and progress to blindness. Along with weight reduction, acetazolamide, which reduces the production of cerebrospinal fluid (CSF), is prescribed as a first-line treatment. Its efficacy is inconsistent in resolving papillary edema and there are many side effects.

In the event of ineffectiveness or dependence on acetazolamide associated with hygiene and dietetic rules, a second line of therapy is then considered: neurosurgical (internal shunt of the LCS) or endovascular (venous stenting) treatment.

These invasive techniques have each proven their effectiveness in the rapid and permanent resorption of OP, allowing improvement or preservation of visual function. In terms of induced morbidity, the superiority of one technique over the other, if it exists, has not been established.

Our objective is to compare the efficacy, safety, and safety of LCS bypass surgery versus venous sinus stenting in HTICi with moderate to severe visual impairment after failure of medical treatment defined by the absence of resorption of the OP after several months

DETAILED DESCRIPTION:
Intervention 1 Name : internal ventricular shunt (neurosurgery)

Other name [facultatif] :

Description :

The internal ventricular shunt consists of the introduction of a catheter from a lateral ventricle into the atrium or peritoneum. It is associated with a valve whose opening pressure is adjustable. The goal is that cerebrospinal fluid can be absorbed extra-cranial.

Intervention 2 Name : endovacascular stenting (interventional neuroradiology)

Other name [facultatif] :

Description :

The placement of a vascular endoprosthesis (stent) is an interventional neuroradiology procedure aimed, by venous approach (percutaneous puncture), to restore the diameter of a venous sinus. It requires 6 months of antiplatelet aggregation. The aim is to allow better venous drainage from the brain to increase the absorption of cerebrospinal fluid.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 or over
* HTICi proven greater than 25cm of water
* Presence of papillary edema (grade> 0 on the Frisen scale)
* Stenosis of at least one transverse sinus on MRI
* Failure of medical treatment and surgical / interventional indication defined by the medical team taking care of the patient
* Consent to participate in the study

Exclusion Criteria:

* Fulminant HTICi
* Contraindication to antiplatelet aggregation
* Contraindication to one or the other of the interventions under study
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Estimated)
Dates: Start 2022-03-02 (Actual); Primary Completion 2026-03-09 (Estimated); Study Completion 2026-12-07 (Estimated)

PRIMARY OUTCOMES:
Resolution of the papillary edema | 3 months after the procedure
  Resolution of the papillary edema at 3 months defined by: disappearance of the edema (grade 0 on the Frisén scale) or reduction of at least 2 grades of the edema compared to baseline without deterioration of the visual field (Humphrey).

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Bourdillon, MD, Principal Investigator — Fondation A. de Rothschild
Locations (1):
- Fondation A De Rothschild, Paris, Paris, France